CLINICAL TRIAL: NCT07147530
Title: Study to Verify Effectiveness and Safety of the Electrically Powered Orthopedic Exercise Device on Gait Ability in Patients With Hip Joint Diseases: Investigator Initiated, Single Center, Single Group Clinical Trial
Brief Title: Effectiveness and Safety of the Electrically Powered Orthopedic Exercise Device on Gait Ability in Patients With Hip Joint Diseases
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9-2025-0018
Record Dates: First submitted 2025-04-21; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Hip Disease
Keywords: Rehabilitation; Gait; Wearable robot; Hip joint disease

STUDY DESIGN:
Intervention Model Description: Researchers will compare non-wearing and wearing conditions of the electrically powered orthopedic exercise device walking speeds, spatiotemporal parameters, balance in participants and does not establish a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearing conditions of Electrically Powered Orthopedic Exercise Device (Experimental): Participants will undergo gait and balance function tests under both non-wearing and wearing conditions of the electrically powered orthopedic exercise device
  Interventions: Device: Electrically Powered Orthopedic Exercise Device

INTERVENTIONS:
Device: Electrically Powered Orthopedic Exercise Device — Participants who pass the screening undergo an evaluation of gait function and balance ability without wearing the Electrically Powered Orthopedic Exercise Device. Afterward, the patient wears the motorized orthopedic exercise device for a total of four adaptation sessions. In each session, the patient performs short-distance walking within 10 meters while wearing the device to explore the appropriate assistive mode and level of support that match their physical condition. No evaluations are conducted while wearing the device during sessions 1, 2, and 3. After the 4th session, an evaluation identical to the one conducted without the device is performed while wearing it, and a satisfaction survey is conducted.

SUMMARY:
Gait is an essential daily activity performed through the complex coordination of the central and peripheral nervous systems and the musculoskeletal system. Gait disorders can negatively affect quality of life, increase the risk of falls, decrease the ability to perform daily activities, and limit physical activity. Various musculoskeletal diseases can cause gait impairment, with hip osteoarthritis and osteonecrosis of the femoral head (ONFH) being the most representative conditions.

Various interventions can be attempted during the early stages of hip joint disease progression. However, improvement in symptoms does not necessarily indicate a halt in disease progression. As the condition advances in most patients, thinning of the full-thickness hip cartilage or collapse of the femoral head occurs, leading to restricted hip range of motion, weakness of the lower limb muscles and functional deterioration, resulting in the need for total hip arthroplasty.

THA offers significant improvements in pain relief and function, regardless of the patient's preoperative status, and can reduce long-term healthcare costs. However, performing THA at an early stage with minimal functional improvement is not recommended. Postoperative complications, such as infections, aseptic loosening, and instability, are potential risks, with younger patients aged 45-64 showing higher revision surgery rates compared to those aged 65 and older. This highlights the need for new interventions that can delay the time to surgery while improving gait function and muscle strength.

Therefore, this study aims to explore the clinical feasibility of the Angel Suit H10 (Angelrobotics, Seoul, Korea) by assessing whether wearing the Electrically Powered Orthopedic Exercise Device improves gait function in patients with hip joint diseases, along with evaluating user satisfaction and device safety.

DETAILED DESCRIPTION:
(1) Overview of study design This investigator-initiated exploratory study is a pilot study designed to evaluate the effectiveness and safety of the Electrically Powered Orthopedic Exercise Device by measuring and analyzing gait function and balance ability in patients with hip joint diseases under both non-wearing and wearing conditions.

(2) Experimental Group and Evaluation Procedures

1. Participant Selection:

   This study includes a single test group with a total of 30 participants. The selection of participants for the electrically powered orthopedic exercise device and the overall study process will be conducted under the prescription and guidance of a rehabilitation medicine specialist, and supervised by assistants (physicians and occupational therapists). The examiner will collect clinical information and conduct a screening assessment for each participant.
2. Evaluation Phase Without Device:

   After the screening test, participants undergo assessments of walking ability and balance without wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist).
3. Pre-Adaptation Phase:

   After the evaluations without the device, a total of four adaptation sessions are conducted, during which the participant wears the device and performs short-distance walking within 10 meters. These sessions are designed to help the participant become familiar with the operation and wearing method of the H10 device. Appropriate device settings are configured for each participant to minimize any potential inexperience or anxiety during use. Participants must complete all four adaptation sessions, and each session should be conducted within a two-week interval.
4. Evaluation Phase:

After completing all four adaptation sessions, participants undergo assessments of walking ability and balance while wearing the motorized orthopedic exercise device. A 10-minute rest period is provided between each assessment. If the participant wishes, additional rest time is allowed and recorded in the case report form. The assessments include the 10-Meter Walk Test, the 6-Minute Walk Test, the Timed Up and Go Test, and the Berg Balance Scale. These evaluations are conducted in the rehabilitation function testing room on the second floor of the facility under the supervision of the research team (physician and either a physical or occupational therapist). After the evaluations are completed, a usability and satisfaction survey regarding the motorized orthopedic exercise device is conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 19 or older
2. Individuals diagnosed with hip osteoarthritis of Kellgren-Lawrence (K-L) Grade 1-4
3. Individuals diagnosed with avascular necrosis of the femoral head at Association Research Circulation Osseous(ARCO) Stage 1-4
4. Individuals able to sit at the edge of a bed without assistance and stand for 10 seconds regardless of support
5. Individuals who are Functional Ambulatory Category (FAC) score of 1-3
6. Individuals who visited Yongin Severance Hospital, understood the study, and signed informed consent
7. Individuals who have adequate cognitive ability (Korean Mini-Mental State Examination score ≥ 20)

Exclusion Criteria:

1. Individuals who have contraindications for lower limb weight-bearing such as severe joint contractures, osteoporosis, or untreated fractures
2. Individuals who have progressive or unstable brain diseases or neurological paralysis from stroke
3. Individuals who have active infections or open wounds hindering device use
4. Individuals who have significant leg length discrepancies
5. Individuals who have severe deformities or contractures in the lower extremities
6. Individuals who have history of poliomyelitis
7. Individuals inable to maintain seated or standing positions independently
8. Individuals who have severe spasticity (Modified Ashworth Scale grade ≥ 2)
9. Individuals who have bone metastases from cancer
10. Individuals who have severe internal diseases affecting device use (e.g., cardiovascular or respiratory diseases)
11. Individuals who have cognitive impairments preventing cooperation with device use
12. Individuals who have complaints of device-related side effects or potential rehabilitation discontinuation
13. Patients who are determined to be pregnant or potentially pregnant based on the medical interview
14. Individuals who have any other clinically significant findings deemed inappropriate by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-04-06 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
10-Meter Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk 14 m, including 2 m at both ends for acceleration and deceleration, at their comfortable speed. Gait speed was calculated by dividing the 10m distance by the time taken.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Researchers ask patients to rise from a seated position, walk a distance of 3 m, turn around, return to the chair, and sit back. The average time of three trials was recorded as a result
6-Minute Walk Test | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are instructed to walk back and forth along the 30-meter path as many times as possible within 6 minutes. The examiner records the total distance covered, abnormal gait patterns, and the time of occurrence of any gait deviations.
Berg balance scale (BBS) | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  Patients are asked to perform 14 tasks regarding the static and dynamic balance of patients. Each task was rated on a five-point scale from 0 to 4, with a total score of 56.
Spatiotemporal Parameters of Gait : Total Step Count | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Total Step Count: The total number of steps taken during walking.
Spatiotemporal Parameters of Gait : Cadence | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Cadence: The number of steps taken per minute, measured in steps per minute (spm).
Spatiotemporal Parameters of Gait : Self-Selected Walking Speed | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Self-Selected Walking Speed: The participant's walking speed when walking naturally at a comfortable pace.
Spatiotemporal Parameters of Gait : Distance | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Distance: The total distance covered during walking, measured in meters (m).
Spatiotemporal Parameters of Gait : Stride Length | A baseline assessment without wearing the device will be conducted on the same day as session 1, and an end-point assessment while wearing the device will be conducted on the same day as session 4
  While the participant performs the test wearing an insole-type gait analyzer, spatiotemporal gait parameters are collected and recorded.
  Stride Length: The distance between the heel of one foot to the heel of the same foot during consecutive steps. Measured in meters (m), stride length is adjusted for height to account for differences in body size.
Satisfaction evaluation | Upon completion of the end-point assessment conducted on the same day as session 4
  Participants will complete a satisfaction survey for usability and satisfaction assessment of the electrically powered orthopedic exercise device, based on the Korean version of the Quebec User Evaluation of Satisfaction with assistive Technology (K-QUEST 2.0).21 This survey consists of 12 items on a 5-point scale. Participants rate their satisfaction with the assistive device and related services

CONTACTS AND LOCATIONS:
Overall Officials: Na Young Kim, MD, PhD, Principal Investigator — Severance Hospital
Locations (1):
- Yongin Severance Hospital, Yongin-si, Gyeonggi-do, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther. 2013 Feb;93(2):158-67. doi: 10.2522/ptj.20120171. Epub 2012 Sep 27. PMID 23023812
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Hwang R, Morris NR, Mandrusiak A, Mudge A, Suna J, Adsett J, Russell T. Timed Up and Go Test: A Reliable and Valid Test in Patients With Chronic Heart Failure. J Card Fail. 2016 Aug;22(8):646-50. doi: 10.1016/j.cardfail.2015.09.018. Epub 2015 Oct 9. PMID 26456063
- [Background] Santos M, Zdravevski E, Albuquerque C, Coelho PJ, Pires IM. Ten Meter Walk Test for motor function assessment with technological devices based on lower members' movements: A systematic review. Comput Biol Med. 2025 Mar;187:109734. doi: 10.1016/j.compbiomed.2025.109734. Epub 2025 Feb 3. PMID 39904103
- [Background] Dolny DG, Collins MG, Wilson T, Germann ML, Davis HP. Validity of lower extremity strength and power utilizing a new closed chain dynamometer. Med Sci Sports Exerc. 2001 Jan;33(1):171-5. doi: 10.1097/00005768-200101000-00026. PMID 11194105
- [Background] Kim Heon-tae, Moon Jun-bae, Ryu Seung-ho, and Kang Min-soo. Validity study of the Korean version of the International Physical Activity Questionnaire (IPAQ): Verification of construct-related validity. Korean Journal of Physical Education No. 2017;56
- [Background] Gajdosik RL, Bohannon RW. Clinical measurement of range of motion. Review of goniometry emphasizing reliability and validity. Phys Ther. 1987 Dec;67(12):1867-72. doi: 10.1093/ptj/67.12.1867. PMID 3685114
- [Background] Cuthbert SC, Goodheart GJ Jr. On the reliability and validity of manual muscle testing: a literature review. Chiropr Osteopat. 2007 Mar 6;15:4. doi: 10.1186/1746-1340-15-4. PMID 17341308
- [Background] Mehrholz J, Wagner K, Rutte K, Meissner D, Pohl M. Predictive validity and responsiveness of the functional ambulation category in hemiparetic patients after stroke. Arch Phys Med Rehabil. 2007 Oct;88(10):1314-9. doi: 10.1016/j.apmr.2007.06.764. PMID 17908575
- [Background] Setoguchi D, Kinoshita K, Kamada S, Sakamoto T, Kise N, Kotani N, Goto K, Shiota E, Inoue T, Yamamoto T. Hybrid Assistive Limb improves restricted hip extension after total hip arthroplasty. Assist Technol. 2022 Jan 2;34(1):112-120. doi: 10.1080/10400435.2020.1712498. Epub 2020 Jan 22. PMID 31909703
- [Background] Li J, Wu T, Xu Z, Gu X. A pilot study of post-total knee replacement gait rehabilitation using lower limbs robot-assisted training system. Eur J Orthop Surg Traumatol. 2014 Feb;24(2):203-8. doi: 10.1007/s00590-012-1159-9. Epub 2013 Jan 9. PMID 23412304
- [Background] Rohner E, Mayfarth A, Sternitzke C, Layher F, Scheidig A, Gross HM, Matziolis G, Bohle S, Sander K. Mobile Robot-Based Gait Training after Total Hip Arthroplasty (THA) Improves Walking in Biomechanical Gait Analysis. J Clin Med. 2021 May 29;10(11):2416. doi: 10.3390/jcm10112416. PMID 34072524
- [Background] Koseki K, Mutsuzaki H, Yoshikawa K, Iwai K, Hashizume Y, Nakazawa R, Kohno Y. Early Recovery of Walking Ability in Patients After Total Knee Arthroplasty Using a Hip-Wearable Exoskeleton Robot: A Case-Controlled Clinical Trial. Geriatr Orthop Surg Rehabil. 2021 Jun 28;12:21514593211027675. doi: 10.1177/21514593211027675. eCollection 2021. PMID 34262793
- [Background] Kirkley A, Webster-Bogaert S, Litchfield R, Amendola A, MacDonald S, McCalden R, Fowler P. The effect of bracing on varus gonarthrosis. J Bone Joint Surg Am. 1999 Apr;81(4):539-48. doi: 10.2106/00004623-199904000-00012. PMID 10225800
- [Background] Pham T, Maillefert JF, Hudry C, Kieffert P, Bourgeois P, Lechevalier D, Dougados M. Laterally elevated wedged insoles in the treatment of medial knee osteoarthritis. A two-year prospective randomized controlled study. Osteoarthritis Cartilage. 2004 Jan;12(1):46-55. doi: 10.1016/j.joca.2003.08.011. PMID 14697682
- [Background] Brouwer RW, Jakma TS, Verhagen AP, Verhaar JA, Bierma-Zeinstra SM. Braces and orthoses for treating osteoarthritis of the knee. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD004020. doi: 10.1002/14651858.CD004020.pub2. PMID 15674927
- [Background] Van der Esch M, Heijmans M, Dekker J. Factors contributing to possession and use of walking aids among persons with rheumatoid arthritis and osteoarthritis. Arthritis Rheum. 2003 Dec 15;49(6):838-42. doi: 10.1002/art.11463. PMID 14673971
- [Background] Rajaee SS, Campbell JC, Mirocha J, Paiement GD. Increasing Burden of Total Hip Arthroplasty Revisions in Patients Between 45 and 64 Years of Age. J Bone Joint Surg Am. 2018 Mar 21;100(6):449-458. doi: 10.2106/JBJS.17.00470. PMID 29557860
- [Background] Berliner JL, Brodke DJ, Chan V, SooHoo NF, Bozic KJ. John Charnley Award: Preoperative Patient-reported Outcome Measures Predict Clinically Meaningful Improvement in Function After THA. Clin Orthop Relat Res. 2016 Feb;474(2):321-9. doi: 10.1007/s11999-015-4350-6. PMID 26201420
- [Background] Hawker GA, Badley EM, Croxford R, Coyte PC, Glazier RH, Guan J, Harvey BJ, Williams JI, Wright JG. A population-based nested case-control study of the costs of hip and knee replacement surgery. Med Care. 2009 Jul;47(7):732-41. doi: 10.1097/MLR.0b013e3181934553. PMID 19536034
- [Background] Judge A, Arden NK, Batra RN, Thomas G, Beard D, Javaid MK, Cooper C, Murray D; Exeter Primary Outcomes Study (EPOS) group. The association of patient characteristics and surgical variables on symptoms of pain and function over 5 years following primary hip-replacement surgery: a prospective cohort study. BMJ Open. 2013 Mar 1;3(3):e002453. doi: 10.1136/bmjopen-2012-002453. PMID 23457332
- [Background] Kinds MB, Welsing PM, Vignon EP, Bijlsma JW, Viergever MA, Marijnissen AC, Lafeber FP. A systematic review of the association between radiographic and clinical osteoarthritis of hip and knee. Osteoarthritis Cartilage. 2011 Jul;19(7):768-78. doi: 10.1016/j.joca.2011.01.015. Epub 2011 Jan 31. PMID 21281726
- [Background] Murphy NJ, Eyles JP, Hunter DJ. Hip Osteoarthritis: Etiopathogenesis and Implications for Management. Adv Ther. 2016 Nov;33(11):1921-1946. doi: 10.1007/s12325-016-0409-3. Epub 2016 Sep 26. PMID 27671326
- [Background] Alves EM, Angrisani AT, Santiago MB. The use of extracorporeal shock waves in the treatment of osteonecrosis of the femoral head: a systematic review. Clin Rheumatol. 2009 Nov;28(11):1247-51. doi: 10.1007/s10067-009-1231-y. Epub 2009 Jul 17. PMID 19609482
- [Background] Bennell KL, Buchbinder R, Hinman RS. Physical therapies in the management of osteoarthritis: current state of the evidence. Curr Opin Rheumatol. 2015 May;27(3):304-11. doi: 10.1097/BOR.0000000000000160. PMID 25775185
- [Background] Gay C, Chabaud A, Guilley E, Coudeyre E. Educating patients about the benefits of physical activity and exercise for their hip and knee osteoarthritis. Systematic literature review. Ann Phys Rehabil Med. 2016 Jun;59(3):174-183. doi: 10.1016/j.rehab.2016.02.005. Epub 2016 Apr 1. PMID 27053003
- [Background] Paans N, van den Akker-Scheek I, Dilling RG, Bos M, van der Meer K, Bulstra SK, Stevens M. Effect of exercise and weight loss in people who have hip osteoarthritis and are overweight or obese: a prospective cohort study. Phys Ther. 2013 Feb;93(2):137-46. doi: 10.2522/ptj.20110418. Epub 2012 Sep 27. PMID 23023813
- [Background] Moya-Angeler J, Gianakos AL, Villa JC, Ni A, Lane JM. Current concepts on osteonecrosis of the femoral head. World J Orthop. 2015 Sep 18;6(8):590-601. doi: 10.5312/wjo.v6.i8.590. eCollection 2015 Sep 18. PMID 26396935
- [Background] Joo YB, Sung YK, Shim JS, Kim JH, Lee EK, Lee HS, Bae SC. Prevalence, incidence, and associated factors of avascular necrosis in Korean patients with systemic lupus erythematosus: a nationwide epidemiologic study. Rheumatol Int. 2015 May;35(5):879-86. doi: 10.1007/s00296-014-3147-3. Epub 2014 Oct 10. PMID 25300729
- [Background] Culliford DJ, Maskell J, Kiran A, Judge A, Javaid MK, Cooper C, Arden NK. The lifetime risk of total hip and knee arthroplasty: results from the UK general practice research database. Osteoarthritis Cartilage. 2012 Jun;20(6):519-24. doi: 10.1016/j.joca.2012.02.636. Epub 2012 Mar 3. PMID 22395038
- [Background] Murphy LB, Helmick CG, Schwartz TA, Renner JB, Tudor G, Koch GG, Dragomir AD, Kalsbeek WD, Luta G, Jordan JM. One in four people may develop symptomatic hip osteoarthritis in his or her lifetime. Osteoarthritis Cartilage. 2010 Nov;18(11):1372-9. doi: 10.1016/j.joca.2010.08.005. Epub 2010 Aug 14. PMID 20713163
- [Background] Helmick CG, Felson DT, Lawrence RC, Gabriel S, Hirsch R, Kwoh CK, Liang MH, Kremers HM, Mayes MD, Merkel PA, Pillemer SR, Reveille JD, Stone JH; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part I. Arthritis Rheum. 2008 Jan;58(1):15-25. doi: 10.1002/art.23177. PMID 18163481
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Alexander NB. Gait disorders in older adults. J Am Geriatr Soc. 1996 Apr;44(4):434-51. doi: 10.1111/j.1532-5415.1996.tb06417.x. No abstract available. PMID 8636592
- [Background] Baker JM. Gait Disorders. Am J Med. 2018 Jun;131(6):602-607. doi: 10.1016/j.amjmed.2017.11.051. Epub 2017 Dec 27. PMID 29288631
- [Background] Mirelman A, Shema S, Maidan I, Hausdorff JM. Gait. Handb Clin Neurol. 2018;159:119-134. doi: 10.1016/B978-0-444-63916-5.00007-0. PMID 30482309
- [Background] Kang Y, NA D-L, Hahn S. A validity study on the Korean Mini-Mental State Examination (K-MMSE) in dementia patients. Journal of the Korean neurological association 1997:300-308
- [Background] Lee, Sang-Heon, Bong-Keun Jung, and So-Yeon Park. "Korean Translation and Psychometric Properties of Quebec User Evaluation of Satisfaction Assistive Technology 2.0." Journal of the Korea Academia-Industrial Cooperation Society. The Korea Academia-Industrial Cooperation Society, July 31, 2013.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT07147530/Prot_SAP_000.pdf